CLINICAL TRIAL: NCT01675466
Title: First Laparoscopy or Active Observation in Acute Non-specific Abdominal Pain: The FLO Trial
Brief Title: Study Comparing Early Laparoscopy With Active Observation in Acute Non-specific Abdominal Pain
Acronym: FLO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Professor, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC123
Record Dates: First submitted 2012-07-20; First posted 2012-08-30 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Non-specific Abdominal Pain
Keywords: non-specific abdominal pain; undifferentiated abdominal pain; appendicitis; appendicectomy; appendectomy; surgery; laparoscopy; antibiotics; randomised controlled trial; randomized controlled trial; controlled clinical trial; randomised; placebo
MeSH Terms: conditions — Appendicitis | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early laparoscopy (Active Comparator): early laparoscopy, aiming to achieve this within 12 hours
  Interventions: Procedure: early laparoscopy; Procedure: General anaesthesia; Device: Laparoscopic instruments
- active observation (Placebo Comparator): standard management - the "wait and see" approach with serial examinations and investigations as deemed necessary

INTERVENTIONS:
Procedure: early laparoscopy — Laparoscopy under performed by the surgeon on duty or his/her deputy. The aim is to achieve this within 12 hours of randomisation. This will be performed under general anaesthetic and involve the necessary drugs. The procedure will require laparoscopy instruments. There will be a umbilical port which will be 10mm in size and one 5mm port below this. If pathology is found, a further port will be needed to perform treatment.
  Arms: early laparoscopy
Procedure: General anaesthesia
  Arms: early laparoscopy
Device: Laparoscopic instruments
  Other Names: Laparoscopic camera; Maryland laparoscopic grasper; Endoclinch laparoscopic grasper; Endobag; Laparoscopic suction
  Arms: early laparoscopy

SUMMARY:
Patients with acute abdominal pain comprise a significant proportion of attendances at emergency departments. These patients account for about a third of general surgical admissions in a typical day. In some cases, the diagnosis is clear from baseline investigations (for example in cases of pancreatitis). In other cases, the diagnosis remains unclear but there are signs that necessitate urgent surgery (for example in cases of appendicitis). A final group exists where no clear explanation for the pain is found and where there are insufficient clinical signs to warrant surgery. These patients are said to have "non specific abdominal pain" (NSAP) and present a management dilemma.

Traditionally such patients are managed with a strategy of active observation. Patients are examined at regular intervals and may undergo imaging. In some cases, symptoms and signs progress and surgery is needed while in other cases resolution may occur or a diagnosis may be reached non-operatively allowing focused medical treatment. Recently, two alternative strategies have emerged. Early cross-sectional imaging using CT scanning may identify conditions whilst being non-invasive. This would allow diagnosis and treatment would follow. The alternative strategy of early laparoscopy (key hole surgery) offers the possibility of concomitant therapy, but is invasive.

The study hypothesis is that in patients with acute non-specific abdominal pain active management with laparoscopy on admission will reduce hospital stay and costs when compared to traditional active observation, without increasing complications.

DETAILED DESCRIPTION:
Patients referred to the general surgical service will initially be managed as per routine practice. They will be assessed by a member of the surgical house-staff, simple baseline investigations (full blood count, serum amylase, C-reactive protein, plain radiography) will be requested. Patients will then be reviewed by a registrar or consultant. At this point, a proportion of patients will have clear indications for surgery e.g. free gas on an erect chest x-ray or peritonitis. A further subgroup will be more appropriately managed by further tests on an out-patient basis and these patients will be allowed home. Some patients will have a clear diagnosis e.g. pancreatitis. Patients in each of these groups will be managed according to the usual practice of the responsible consultant surgeon.

There is a final subgroup of patients who are the population of interest for this trial. These are patients in whom no clear diagnosis or safe decision to operate or discharge is possible. Such patients are usually admitted for a period of observation with further investigations or interventions ordered as their clinical picture evolves.

These patients will then be randomly assigned to one of two management options: an active observation arm (control) or early laparoscopy arm.

Active Observation: Patients randomised to this group will receive routine practice and will serve as the trial control group. They will be reviewed regularly by the responsible surgical team. Further investigations and interventions will be requested at the discretion of the responsible team.

Early laparoscopy: Patients randomised to this group will be listed for a diagnostic laparoscopy in the emergency theatre . The aim will be to undertake this procedure within 12 hours of randomisation. The procedure will be performed by the duty consultant surgeon or his / her nominated deputy as is usual practice. Findings at laparoscopy which require surgical intervention e.g. appendicitis will be treated as part of the same procedure as is routine clinical practice.

Follow-up: Each patient will be followed-up on a daily basis by a member of the trial team whilst an in-patient. Complications, further investigations and interventions, unplanned critical care admissions, death, length of hospital stay and final discharge diagnosis will all be recorded. Following discharge, each patient will be reviewed at four weeks and six months. SF36 questionnaires will be completed at each of these visits. In addition, the Hospital In-patient Episode database will be interrogated for further admissions to other hospitals within six months of randomisation

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18
* admission with abdominal pain for up to one week prior to admission deemed to be non-specific pain by senior surgical team member
* patient willing to give full informed consent for participation

Exclusion Criteria:

* patients less than 18 years of age
* pain of greater than 7 days duration
* admission with abdominal pain in previous 6 months
* history of inflammatory bowel disease
* previous history of appendicectomy
* previous surgery rendering laparoscopy unsafe eg. multiple laparotomies
* history of intra-abdominal transplant including retroperitoneal renal allografting
* clinical picture necessitating immediate surgical procedure
* cases involving trauma
* patients who are unable or unwilling to give full informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | the length of inpatient stay
  The primary outcome is the length of inpatient hospital stay which will an expected average of 3 days.

SECONDARY OUTCOMES:
Complications within 30 days | within 30 days following randomisation
  Includes any complication encountered by participants in either arm of the trial in the first 30 days following randomisation.
further radiological investigations during inpatient stay | during inpatient stay
  A secondary outcome measure is the number of radiological tests patients undergo during their inpatient stay following randomisation. These could be ultrasound, plain radiography, CT scanning, MRI scanning. Average inpatient stay is expected to be 3days.
readmission to hospital with abdominal pain | from randomisation to 6 months
SF36 score at 4 weeks | from randomisation to4 weeks
  The Short Form (36) Health Survey is a validated survey of patient health
SF36 score at 6 months | 6 months following randomisation
  The Short Form (36) Health Survey is a validated survey of patient health
upstaging to more severe diagnosis within 6 months | from randomisation to 6 months
further blood investigations during inpatient stay | during inpatient stay
  This refers to the number of further investigations during hospital stay. Average length of stay is expected to be 3 days
further urine tests during inpatient stay | during inpatient stay
  This refers to further urine tests during hospital stay. The average hospital stay is expected to be 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Donagh A Healy, MB, Principal Investigator; Stewart R Walsh, MB MCh, Principal Investigator
Locations (1):
- University Hospital Limerick, Limerick, Limerick, Ireland